CLINICAL TRIAL: NCT05094752
Title: Assessment of the Effects of Early Proprioceptive Stimulations in Patients With Spinal Cord Injury : a Randomized Controlled Trial
Brief Title: Assessment of the Effects of Early Proprioceptive Stimulations in Patients With Spinal Cord Injury
Acronym: Tetra-Mouv
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-A02015-34
Record Dates: First submitted 2021-09-22; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injuries; quadriplegia; proprioceptive stimulation; vibration; spasticity; intensive care units
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Vibration treatment will last eight weeks for each patient, with 4 sessions per week, 30 minutes per session. Subjects of the intervention group will receive proprioceptive stimulations set to create illusions of movement.
  Interventions: Device: Proprioceptive stimulations
- Control group (Sham Comparator): Vibration treatment will last eight weeks for each patient, with 4 sessions per week, 30 minutes per session. Subjects of the control group will receive sham stimulations.
  Interventions: Device: Sham stimulations

INTERVENTIONS:
Device: Proprioceptive stimulations — Vibration treatment will last eight weeks for each patient, with 4 sessions per week, 30 minutes per session. Subjects of the intervention group will receive proprioceptive stimulations set to create illusions of movement.
  Arms: Intervention group
Device: Sham stimulations — Vibration treatment will last eight weeks for each patient, with 4 sessions per week, 30 minutes per session. Subjects of the control group will receive sham stimulations.
  Arms: Control group

SUMMARY:
"Spinal cord injury (SCI) is a dramatic event resulting in a long-term handicap. Appropriate care from admission to the intensive care unit (ICU) is a key element not only for the survival of these patients but also to promote their recovery. Moreover, the studies on natural history of SCI have shown that most of the recovery occurs within the first 3 to 6 months post-injury. This period is therefore crucial for these patients. However, the environment of the ICU and the acute condition of the patients limit the rehabilitation possibilities. In such a context, functional proprioceptive stimulations (Vibramoov™ system, Techno Concept, France) could be a tool of interest.

By using tendon vibrations, the Vibramoov™ system allows to reproduce the proprioceptive signatures of cyclic movements such as walking. Some studies have already demonstrated the benefits of proprioceptive vibrations. However, so far, these benefits have only been studied at the chronic stage of neurological diseases.

The investigators hypothesized that early functional proprioceptive stimulations (FPS) may reduce spasticity and promote sensorimotor recovery in tetraplegic and high paraplegic patients.

To test their hypothesis, the investigators conduct a randomized controlled trial on 40 patients with traumatic SCI. These patients will be stratified into two groups according to the completeness of their lesion. Every patient will be included within ten days post-injury and receive either FPS, either sham stimulations to the joints of the lower limbs, 4 times a week during 8 weeks. the primary outcome measures will assess spasticity. the investigators also assess sensorimotor recovery, pain, muscle wasting, cognitive impairment and functional status. "

ELIGIBILITY:
Inclusion Criteria:

* • Traumatic Spinal Cord Injury at or above level T6

  * Age ≥ 18 years old
  * No pregnancy
  * Not being under guardianship
  * Be affiliated to the French social security system

Exclusion Criteria:

* Orthopedic lesions or any medical condition that prevent the implementation of the protocol within ten days post-injury
* Severe brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Changes in the modified Ashworth scale (MAS) | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  The MAS enables to assess spasticity. The muscle whose spasticity will be assessed are the soleus, gastrocnemius, knee extensors, knee flexors, adductors and gracilis (Score range from 0 to 5 per muscle, higher values represent a higher severity of spasticity)
Changes in the angles of the muscle reaction in the modified Tardieu scale (MTS) | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  The MTS enables to assess the severity of spasticity. The muscle whose spasticity will be assessed are the soleus, gastrocnemius, knee extensors, knee flexors, adductors and gracilis (The outcome is reported in degree, from 0 to 180 degrees, higher values represent a higher dynamic component of spasticity)
Changes in the quality of the muscle reaction in the modified Tardieu scale (MTS) | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  The muscle whose spasticity will be assessed are the soleus, gastrocnemius, knee extensors, knee flexors, adductors and gracilis (Score range from 0 to 5 per muscle, higher values represent a higher severity of spasticity)
Changes in the Spinal cord assessment tool for spastic reflexes (SCATS) | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  This score enables to asses global spasticity (Score range from 0 to 18, higher values represent a higher degree of spasticity)

SECONDARY OUTCOMES:
Changes in the visual analog scale for the auto-assessment of problematic spasticity | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  Score range from 0 to 100, higher values represent a higher degree of problematic spasticity.
Changes in the visual analog scale for the auto-assessment of pain | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury
  Score range from 0 to 100, higher values represent a higher intensity of pain.
Changes in the International standards for neurological classification of spinal cord injury (ISNCSCI) score | At inclusion, and at one week, one month, 2 months, 6 months and 1 year after the injury.
  This score enables to assess sensorimotor recovery (Score range from 0 to 324, higher values represent a better outcome)
Changes in the quadriceps muscle thickness | At inclusion, then twice a week during the first month, and at 2 months, 6 months and 1 year after the injury
  "Measured with ultrasound, average of two measures (at the border between the lower third and upper two-thirds between the anterior superior iliac spine and the upper pole of the patella, and at the midpoint between the anterior superior iliac spine and the upper pole of the patella) (Measure in centimeters, higher values represent a better outcome)"
Changes in the nitrogen balance, | Every 48 hours during the first two weeks, and then once a week for six weeks
  Marker of protein losses (Measure in mmol/L, lower values represent a better outcome)
Number of days between the SCI and the verticalization at 45° | Verticalization is attempted progressively 3 times a week during the 8 weeks of treatment.
  The attempt is successful if the position is maintained for 5 minutes without adverse effect. The verticalization protocol will remain the same as the one commonly used in the ICU. According to this protocol, verticalization will be progressive and mean blood pressure will be monitored continuously. The attempt is stopped if the patient feels unwell (signs of intolerance) or if the mean blood pressure drops by more than 20% (Measure in days, higher values represent a lower outcome)
Number of days between the SCI and the verticalization at 70° | Verticalization is attempted progressively 3 times a week during the 8 weeks of treatment.
  The attempt is successful if the position is maintained for 5 minutes without adverse effect. The verticalization protocol will remain the same as the one commonly used in the ICU. According to this protocol, verticalization will be progressive and mean blood pressure will be monitored continuously. The attempt is stopped if the patient feels unwell (signs of intolerance) or if the mean blood pressure drops by more than 20% (Measure in days, higher values represent a lower outcome)
Changes in the Spinal cord independence measure (SCIM) | At 2 months, 6 months and 1 year after the injury
  This measure enables to assess functional status (Score range from 0 to 100, higher values represent a better outcome)
Changes in the Montreal cognitive assessment (MoCA) | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Score range from 0 to 30, higher values represent a better outcome)
Changes in the time to complete the bells cancellation test to assess cognitive impairments | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Measure in minutes and seconds, lower values represent a better outcome)
Changes in the number of omissions in the bells cancellation test to assess cognitive impairments | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Lower values represent a better outcome)
Changes in the digit span test to assess cognitive impairments | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Higher values represent a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard VIGUE, Principal Investigator — APHP
Locations (1):
- Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinache F, de Crouy AC, Boutin A, Duranteau J, Vigue B. Early functional proprioceptive stimulation in high spinal cord injury: a pilot study. Front Rehabil Sci. 2025 Feb 26;6:1490904. doi: 10.3389/fresc.2025.1490904. eCollection 2025. PMID 40078600